CLINICAL TRIAL: NCT02473783
Title: An I-123-ADAM SPECT Imaging Study to Evaluate the Serotonin Transporter (SERT) Availability for Prognosing Major Depressive Disorder (MDD) Treatment and Assisting in Detecting MDD
Brief Title: The Serotonin Transporter Availability for Prognosing Major Depressive Disorder (MDD) Treatment and Detecting MDD
Acronym: STAPMDDTDM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: National Atomic Research Institute, Taiwan (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Director of Department of Psychiatry, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INEI-1A20090409
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): The subjects with major depressive disorder who are screened into this study were scheduled for T1-weighted MRI (MRI examination results within 6 months before study are acceptable) prior to the visit of SPECT scans to confirm the absence of organic lesion in the brain and to co-register with SPECT images for the delineation of brain anatomical locations. After the screening visit, eligible subjects received I-123-ADAM SPECT before and after the pharmacological intervention with Sertraline HCl for a treatment period of six weeks. The subjects were observed until no clinically significant adverse events at the drug administration visits before being dismissed.
  Interventions: Drug: Sertraline HCl; Other: I-123-ADAM SPECT

INTERVENTIONS:
Drug: Sertraline HCl — The regimen of Sertraline HCl will be administered with starting dose from minimum 25 mg/day for 1 week and maintenance dose of at least 50 mg/day up to 200 mg/day for the rest of 5 weeks.
  Other Names: Zoloft
Other: I-123-ADAM SPECT — The subjects underwent the SPECT scan after I-123-ADAM (185 MBq, 5mCi) IV injection.

SUMMARY:
Objectives:

1. To evaluate the relationship between improvement of Hamilton Depression Rating Scale (HAMD) score and basal SERT availability (binding potential) for the prognosis of MDD subjects being treated with Sertraline HCl
2. To evaluate the SERT availability by means of I-123-ADAM SPECT imaging study for assisting in detecting MDD
3. To evaluate the relationship between basal HAMD score and basal SERT availability for MDD subjects
4. To evaluate the relationship between basal HAMD somatic subscale score and basal SERT availability for MDD subjects
5. To evaluate the relationship between change of SERT availability and change of HAMD score for MDD patients being treated with Sertraline HCl

DETAILED DESCRIPTION:
Background:

Serotonin transporter (SERT) plays an important role in the pathophysiology of psychiatric disorders such as anxiety and depression and is the primary target of the selective serotonin reuptake inhibitors (SSRIs) which are posited to exert their effect in treating psychiatric disorders aforementioned by this mechanism. I-123-ADAM is a selective radioligand for imaging SERT using SPECT. Research showed that it displayed an extremely high binding affinity to SERT sites. Previous literature also suggested the potential role of I-123-ADAM SPECT as useful in understanding how serotonin system affected depression. This study aims to evaluate the SERT availability by means of I-123-ADAM SPECT imaging study in drug-free subjects for prognosing MDD treatment and assisting in detecting MDD.

Methods:

We enrolled patients who had major depressive disorder but was free from prior antidepressant medication for at least 5 times of elimination half-lives and healthy controls. The patients with major depressive disorder (N=20) received I-123-ADAM SPECT before and after the pharmacological intervention with Sertraline HCl for a treatment period of six weeks. All healthy subjects (N=17) had only basal I-123-ADAM SPECT. The relationship between improvement of depressive symptoms and basal SERT availability for the prognosis of MDD subjects being treated with Sertraline HCl will be analyzed. In addition, the association between the efficacy of treatment with Sertraline HCl and the change of SERT availability will also be investigated. The control group were selected in order to distinguish the difference of basal SERT binding potential of I-123-ADAM between healthy and MDD subjects.

ELIGIBILITY:
Inclusion Criteria:

- For MDD subjects

1. Subject meets the DSM-IV criteria for MDD
2. Subject has a minimum score of 18 on the 17-item HAMD total score
3. Subject has a minimum score of 2 on item 1, depressed mood, of HAMD
4. Subject is free from prior antidepressant medication for at least 5 times of elimination half-lives

For healthy subjects

1. Subject without past or current neuropsychiatric illnesses based on a clinical interview including Mini-International Neuropsychiatric Interview (M.I.N.I.) and a physical examination
2. Subject without exposure to psychotropic medication or other substances known to affect the brain serotonin system within 1 year prior to entering the study

Exclusion Criteria:

1. Subject with history of any co-morbid neuropsychiatric disease
2. Subject with history of treatment resistant to at least two full doses and courses of antidepressant medication
3. Subject with history of alcohol or substance dependence or abuse
4. Subject with allergic history to the investigational products
5. Subject with severe cardiovascular disease or cerebrovascular disease which is judged by investigators for safety concerns as inappropriate for this study
6. Subject with malignancy within past 5 years
7. Subject with any diseases judged by investigators as inappropriate for this study
8. Female subject being pregnant, nursing, or lactating
9. Female subject of childbearing potential not using a medically acceptable form of birth control
10. Subject is unable to undergo MRI scan to confirm the absence of organic lesion in the brain and to co-register with SPECT images for the delineation of brain anatomical locations
11. Subject participated in any investigational drug trial within 4 weeks before entering this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from Oct-07-2011 to Nov-28-2012. The recruitment site was a psychiatric outpatient in a medical center.
Pre-assignment Details: The treatment group:
  No significant events in the study that occur after participant enrollment.
  The healthy control group:
  No significant events in the study that occur after participant enrollment.
Groups:
- Healthy Control Group: All healthy subjects had only basal I-123-ADAM SPECT scanning
Period: Overall Study
Arm/Group | Treatment Group | Healthy Control Group
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treatment group received I-123-ADAM SPECT scanning before and after the pharmacological intervention with Sertraline HCl for a treatment period of six weeks. All healthy subjects had only basal I-123-ADAM SPECT.
Groups:
- Healthy Control Group: All healthy subjects (N=17) had only basal I-123-ADAM SPECT scanning.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Healthy Control Group | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.15 (12.35) | 36.35 (12.72) | 37.32 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 17 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 20 | 17 | 37
Hamilton Depression Rating Scale (HAMD) total score [Mean (Full Range); unit: units on a scale] — The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The patient is rated by a clinician on 17 items scored either on a 3-point or 5-point Likert-type scale. The range of the total score (summed) is from 0 to 52.The higher total score suggests the more severe depression.
  units on a scale | 22.90 [18 to 30] | NA [NA to NA] — We did not measure HAMD scores of Healthy control group. | 22.90 [18 to 30]
serotonin transporter (SERT) binding potential over right basal ganglion [Mean (Standard Deviation); unit: ratio] — Binding potential (BP) is a ratio of specific to non-displaceable binding (BP = (target region (right basal ganglion) - cerebellum) / cerebellum)
  ratio | 0.52 (0.28) | 0.94 (1.32) | 0.68 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: The SERT Binding Potential (BP) --(Only the Treatment Group Was Assessed)
Description: Binding potential (BP) is a ratio of specific to non-displaceable binding (BP = (target region - cerebellum) / cerebellum)
Time Frame: 6 weeks (The Healthy control Group only had the scanning at baseline)
Population: All the participants in the Intention -to-treatment group completed the study. Since the healthy control group did not receive the pharmacological intervention, they underwent only the baseline assessments but not the follow-up ones. Therefore, we reported only the outcome measures of the treatment group.
Measure: Mean (Standard Deviation); unit: a ratio of target region to background
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
a ratio of target region to background | 0.34 (0.26)

2. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) Total Scores
Description: The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. It contains 17 items to be rated. Each item on the questionnaire is scored on a 3 or 5 point scale. The range of the total score (summed) is from 0 to 52.The higher total score suggests the more severe depression.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment Group: The subjects with major depressive disorder were assessed with Hamilton Depression Rating Scale (HAM-D) before and after 6 weeks of Sertraline HCl treatment.
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
units on a scale | 5.25 (4.01)

3. Secondary Outcome: Safety Assessments - the Tolerability of Injection of I-123-ADAM Solution
Description: Pain Scores as measured by the Visual Analog Scale (0-10) for the tolerability of injection of I-123-ADAM solution. Higher values represent a worse outcome.
Time Frame: assessed at -5~0 days and 6 weeks ±5 days, -5~0 days reported (I-123-ADAM SPECT scan)
Population: All the participants in the Intention -to-treatment group completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Healthy Control Group
Number analyzed (Participants) | 20 | 17
units on a scale | 1.52 (2.76) | 0.88 (1.96)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The healthy control group did not receive the pharmacological intervention, they underwent only the baseline assessments and were only monitored for adverse events at baseline.
Arm/Group | Treatment Group | Healthy Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 1/20 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=20) | Healthy Control Group (N=17)
conjunctivitis (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes